CLINICAL TRIAL: NCT01942382
Title: Clinical Pharmacology Study of JNS010 (Paliperidone Palmitate) in Subjects With Schizophrenia
Brief Title: A Clinical Pharmacology Study of JNS010 (Paliperidone Palmitate) in Patients With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100413; PALM-JPN-3 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2013-09-10; First posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; JNS010; Paliperidone Palmitate; Clinical Pharmacology
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Participants will receive 4 injections of paliperidone palmitate 150 milligram in the deltoid muscle on Days 1, 8, 36, and 64.
  Interventions: Drug: Paliperidone palmitate
- Treatment B (Experimental): Participants will receive 4 injections of paliperidone palmitate 75 milligram in the deltoid muscle on Days 1, 8, 36, and 64.
  Interventions: Drug: Paliperidone palmitate
- Treatment C (Experimental): Participants will receive 4 injections of paliperidone palmitate 75 milligram in the gluteal muscle on Days 1, 8, 36, and 64.
  Interventions: Drug: Paliperidone palmitate

INTERVENTIONS:
Drug: Paliperidone palmitate — Participants will receive 4 injections of paliperidone palmitate of concentration ranging from 75 to 150 milligram equivalents in deltoid or gluteal muscle as randomized to treatment group A, B, or C on Days 1, 8, 36, and 64.
  Other Names: JNS010

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (study of what the body does to a drug) and safety of paliperidone palmitate ranging from 75 to 150 milligram equivalents in repeated doses (4 injections) administered in the deltoid muscle (muscle in the shoulder) or gluteal muscle (group of muscles present in the buttocks) in participants with schizophrenia.

DETAILED DESCRIPTION:
This is a multicenter (study conducted at multiple sites), open label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), parallel-group (each group of participants will be treated at the same time) study. Approximately, 60 participants will be enrolled in the study. This study will consist of a screening phase (maximum 14 days), an observation phase (92 days), and a follow-up phase (98 days). Participants will be randomly assigned to treatment group A, B, or C. During the observation phase, participants will receive injections of paliperidone palmitate of concentration ranging from 75 to 150 milligram equivalents in the deltoid muscle or gluteal muscle as applicable on Days 1, 8, 36, and 64 alternating between sides (left/right). Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, vital signs, physical examination, injection site reaction, drug-induced extrapyramidal symptoms scale, and visual analog scale which will be evaluated throughout the study. The total study duration for each participant will be approximately 190 days.

ELIGIBILITY:
Inclusion Criteria:- Participants had to have the capability to provide informed consent in writing to participate in the study

* Participants with a diagnosis of schizophrenia in accordance with the diagnostic criteria for Diagnostic and Statistical Manual of Mental Disorders -IV-TR (DSM-IV-TR)
* Participants whose psychiatric symptom is considered stable by the investigator/subinvestigator at the time of giving informed consent
* Participants with a Positive and Negative Syndrome Scale (PANSS) score of less than or equal to 4 (moderate) in the following 9 items at screening: delusion, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility, uncooperativeness, poor impulse control
* Participants with an experience of taking a risperidone formulation or a paliperidone formulation by 8 days before the initial day (Day 1) of the study treatment

Exclusion Criteria:- DSM-IV-TR diagnosis other than schizophrenia

* DSM-IV-TR diagnosis of substance-related disorders within 180 days before the date of screening
* At a risk of suicide or other-injurious behavior as considered by the investigator/subinvestigator , and participants with a history of suicide attempts
* Concurrent condition of Parkinson's disease (except for drug-induced extrapyramidal syndrome) - Concurrent condition or history of symptomatic cerebrovascular accident

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of unchanged drug (Paliperidone palmitate) | Days 1 to 190
Plasma concentration of active metabolite (paliperidone) | Days 1 to 190
Plasma concentration of enantiomer of paliperidone palmitate (R078543) | Days 1 to 190
Plasma concentration of enantiomer paliperidone palmitate (R078544) | Days 1 to 190
Maximum Observed Plasma Concentration (Cmax) of paliperidone palmitate | Days 1 to 190
  The Plasma Concentration (Cmax) is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of paliperidone palmitate | Days 1 to 190
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of paliperidone palmitate | Days 1 to 190
  The Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) is a measure of the plasma paliperidone concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Number of participants with adverse events | Up to Day 190

SECONDARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Screening, Baseline (Day 1), Days 8, 36, 64, and 92
  The PANSS is a medical scale that assesses various symptoms of schizophrenia. The symptoms are rated on a 7-point scale from 1 (absent) to 7 (extreme psychopathology). The total score is the sum of all 30 PANSS items, with a range of 30 (absent) to 210 (extreme ill). Higher scores indicate worsening.
Change From Baseline in Clinical Global Impression Severity (CGI-S) Scale Score | Screening, Baseline (Day 1), Days 8, 36, 64, and 92
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- See also: Clinical pharmacology study of JNS010 (Paliperidone palmitate) in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2965&filename=CR100413_CSR.pdf